CLINICAL TRIAL: NCT03194308
Title: Safer Conception for Women: PrEP Uptake/Adherence to Reduce Periconception HIV Risk for South African Women
Brief Title: Safer Conception for Women - Understanding Use of Periconception PrEP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); University of Witwatersrand, South Africa (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Lynn T Matthews, Assistant Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2016P001535; 1R01MH108412 (NIH)
Record Dates: First submitted 2017-06-19; First posted 2017-06-21 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: HIV Prevention; Conception
Keywords: HIV risk reduction; Safer Conception; Pre-exposure prophylaxis; South Africa; Women; Reproductive Health

STUDY DESIGN:
Intervention Model Description: All participants are assigned to the Safer Conception study intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- HIV-uninfected women (Other): A sample of 350 HIV-uninfected women who are not currently pregnant, in a stable relationship (≥6 months) with a self-reported infected or unknown serostatus partner and personal or partner plans for pregnancy in the next 12 months. Women will be offered safer conception counseling based on South African guidelines plus daily, oral tenofovir/emtricitabine (TDF/FTC) as pre-exposure prophylaxis (PrEP) during periconception and pregnancy.
  Interventions: Behavioral: PrEP for Safer Conception

INTERVENTIONS:
Behavioral: PrEP for Safer Conception — Evaluation of uptake of and adherence to PrEP and safer conception strategies including: CHCT, ART for the infected partner, and uptake of contraception for those who decide not to conceive by enrolled women, during periconception and pregnancy follow up.

SUMMARY:
Women who choose to conceive with an infected or unknown serostatus partner in HIV-endemic settings need prevention strategies to reduce periconception HIV acquisition risk. Women at high risk for acquiring HIV during pregnancy need risk reduction strategies to protect themselves and their babies. Evaluating uptake of and adherence to antiretrovirals as pre-exposure prophylaxis in this population is crucial to understanding whether and how this novel prevention strategy should be incorporated into HIV-risk reduction packages for at- risk women planning or with pregnancy.

DETAILED DESCRIPTION:
In HIV-endemic settings, many HIV-uninfected women choose to conceive with an HIV-infected or unknown-serostatus partner. For a woman who cannot depend on a partner to test, initiate and adhere to ART, sex without condoms puts her at high risk of acquiring HIV and increases the risk of perinatal transmission to her child. Daily, oral TDF/FTC PrEP dramatically reduces a woman's risk of HIV-acquisition and is the only female-controlled option for reducing the risk of periconception HIV-acquisition. Understanding whether daily, oral PrEP is feasible for uninfected women seeking pregnancy is critical to reducing HIV incidence among women and their children.

Placebo-controlled trials identified adherence as a major challenge to long-term PrEP use. However, women are eager for prevention strategies that allow for conception, and we hypothesize that adherence to a proven prevention strategy, for a limited time with the motivation to have a healthy child, will confer drug levels required to prevent HIV transmission. This project will inform whether daily, oral PrEP is a feasible HIV-prevention strategy for South African women who intend to conceive with risky partners. Given the repercussions of acquiring HIV during conception and pregnancy, this is an important step towards providing a key prevention strategy to women and their children.

ELIGIBILITY:
Inclusion Criteria:

* Female, Aged 18-35 years
* Not pregnant, HIV-uninfected
* Likely to be fertile based on responses to reproductive history assessment
* Not on a long-acting family planning method
* Likely to have a child in the next year, either by response to modified CDC Pregnancy Risk Assessment [2-5]), or meeting the other inclusion criteria.
* With a stable (>= 6 months) partner she reports as HIV-infected or HIV-serostatus unknown, (if >1 desired pregnancy partner, we will ask her to identify the most likely pregnancy partner- based on her own assessment of sexual frequency, fertility, etc.)
* Able to participate in the informed consent process
* Fluent in English or isiZulu

Exclusion Criteria:

* Living at or planning to relocate to a location incompatible with study participation in the next year
* Active drug or alcohol use that, in the opinion of the research study team, would interfere with adherence to study requirements
* Active illness requiring systemic treatment and/or hospitalization within 30 days prior to study entry that in the opinion of the research study team, might otherwise interfere with adherence to study requirements
* Inability to adhere to the study schedule and/or study procedures
* Enrolment in studies which may conflict with their participation in this proposed study.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 330 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2021-07-21 (Actual); Study Completion 2021-07-21 (Actual)

PRIMARY OUTCOMES:
Evaluation of uptake of and adherence to PrEP | minimum of 12 months through pregnancy outcome (maximum 21 months)
  The primary objective will be the evaluation of uptake of (collection of one month's supply) and adherence to PrEP (measured by quarterly plasma tenofovir levels) by women, during periconception and pregnancy follow up.

SECONDARY OUTCOMES:
Safer Conception Strategies | minimum of 12 months through pregnancy outcome (maximum 21 months)
  Secondary outcomes include uptake of safer conception strategies including CHCT, ART for the infected partner, uptake of contraception for those who decide not to conceive; HIV transmission events, infant outcomes, and findings from qualitative interviews to further inform the conceptual framework for periconception PrEP uptake and adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Lynn T Matthews, MD, MPH, Principal Investigator — Mass General Hosptial
Locations (1):
- Maternal, Adolescent, and Child Health Research Unit (MRU), Durban, KwaZulu-Natal, South Africa

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kwach B, Odoyo JB, Lauff AR, Omollo V, Rono B, Ogello V, Mann V, Kwena Z, Thomas K, Sharma M, Morton JF, Ngure K, Bukusi E, Mugwanya KK, PrEP Care Team OS. Evaluating the effectiveness of a One-Stop PrEP Care model to enhance HIV prevention: a protocol for a cluster-randomised trial in Kisumu County, Kenya. BMJ Open. 2025 Sep 8;15(9):e097792. doi: 10.1136/bmjopen-2024-097792. PMID 40921636
- [Derived] Matthews LT, Jaggernath M, Kriel Y, Smith PM, Haberer JE, Baeten JM, Hendrix CW, Ware NC, Moodley P, Pillay M, Bennett K, Bassler J, Psaros C, Hurwitz KE, Bangsberg DR, Smit JA. Oral preexposure prophylaxis uptake, adherence, and persistence during periconception periods among women in South Africa. AIDS. 2024 Jul 15;38(9):1342-1354. doi: 10.1097/QAD.0000000000003925. Epub 2024 May 27. PMID 38752557
- [Derived] Matthews LT, Jaggernath M, Kriel Y, Smith PM, O'Neil K, Haberer JE, Hendrix C, Baeten JM, Ware NC, Wirth K, Psaros C, Bangsberg DR, Smit JA. Protocol for a longitudinal study to evaluate the use of tenofovir-based PrEP for safer conception and pregnancy among women in South Africa. BMJ Open. 2019 Jul 26;9(7):e027227. doi: 10.1136/bmjopen-2018-027227. PMID 31350241